# 研究方案

抗生素联合利福平治疗葡萄球菌假体周围感染的疗效与并发症 ——一项多中心、随机对照试验

# 研究简称

## **CART-PJI**

(Efficacy and Complications of Combining Antibiotics with Rifampin for Treating Staphylococcal Periprosthetic Joint Infection:

A Multicenter Randomized Controlled Trial)

版 本: v2.0

日 期: 2024年10月12日

## 方案签字页

## 研究者声明

我将根据 ICH-GCP 及 CFDA《临床试验质量管理办法》规定,认真履行研究者职责。我已经阅读并了解此研究方案,本项研究将根据《赫尔辛基宣言》和 ICH-GCP 规定的道德、伦理和科学的原则进行;我同意按照本方案设计及规定开展此项目临床研究。我将负责做出与临床相关的医学决定,保证受试者在研究期间出现不良事件时及时采取措施及适当的治疗;我知道正确报告严重不良事件的程序,我将根据要求记录和报告这些事件。我保证将数据准确、完整、及时、合法地记录在病例报告表中。我将接受课题负责单位派遣的监查员或稽查员稽查,确保临床研究的质量。我同意研究结果由课题负责单位在相关专业刊物上发表。我将在研究开始前提供一份履历,呈送伦理委员会。

| 研究单位: |
|--------|
| 研究者签字: |
| 签字日期: |

# 方案摘要

| 研究名称 | 抗生素联合利福平治疗葡萄球菌假体周围感染的疗效与并发症——一项多中心、<br>随机对照试验 |
|---|---|
| 研究目的 | 评价抗生素联合利福平对假体周围感染疗效的影响 |
| 研究设计 | 各个中心符合纳入标准的 PJI 患者,完成 DAIR 或移除假体翻修术后,随机分配至<br>抗生素联合利福平治疗组或单纯抗生素治疗组,统计并分析两组患者的感染控制<br>率及并发症发生率 |
| 课题负责单位 | 福建医科大学附属第一医院 |
| 研究对象 | 各中心人工关节感染接受手术治疗后的患者 |
| 纳入排除标准 | <ol> <li>入选标准 <ol> <li>根据 MSIS 标准确诊为 PJI</li> <li>经微生物培养确定致病菌为葡萄球菌并进行药敏测试</li> <li>有完整临床资料</li> <li>年龄 &lt; 80 周岁,没有严重的合并症或免疫抑制状态</li> <li>患者自愿参与本研究,并在身体与精神上可耐受本研究的治疗过程和各项检测,已签署知情同意书,并通过所有参与本研究的医院伦理委员会审核 </li> <li>排除标准 <ol> <li>术前其他部位有慢性炎症者</li> <li>非葡萄球菌感染或混合感染者</li> <li>患者存在其他可能影响结果的疾病,如免疫缺陷、肝肾功能不全</li> <li>预期寿命小于半年者</li> <li>研究者判断患者因依从性问题不再符合该研究的标准</li> <li>对利福平过敏者</li> </ol> </li> </ol></li></ol> |
| 诊断指标 | 人工关节感染 MSIS 诊断标准(2014 版) |

| | 1. 主要诊断指标(满足以下2条中任意1条): |
|---|---|
| | 1) 存在与假体相通的窦道; |
| | 2)受累人工关节的2处假体周围组织或关节液标本中分离出同一病原体。 |
| | 2. 次要诊断指标 (满足以下 5 条中任意 3 条): |
| | 1) 红细胞沉降率 (ESR>30)或 C 反应蛋白 (CRP>10)水平升高; |
| | 2) 关节液白细胞计数升高 (>3000)或白细胞酯酶试纸条测试结果(++); |
| | 3) 关节液中性粒细胞(PMN)百分比升高 (>80%); |
| | 4)阳性病理表现:400倍放大率下,假体周围组织的病理学分析在5个高倍镜视野下发现>5个中心粒细胞; |
| | 5)假体周围组织或关节液标本中1次培养分离出微生物。 |
| | 主要疗效指标 |
| | 1.感染清除率,感染清除率计算公式:判定为感染清除的受试者例数/完成随访的受试者总例数。感染清除定义为:患者(1)感染根除,伤口愈合,无瘘管、无引流、无痛感,无同一菌种感染复发;(2)无因感染再次手术干预;(3)没有发生 PJI相关疾病如败血症、坏死性筋膜炎等导致的死亡。 |
| 疗效指标 | 2. 与 PJI 相关的不良事件。 |
| | 次要疗效指标 |
| | 1.术后的功能评分; |
| | 2.术后假体松动的比率、翻修率、需要移除假体所占比率; |
| | 3.抗生素并发症的发生率。 |
| 统计学分析 | 包括描述性分析、抗生素方案、手术策略分层分析和抗生素方案与感染清除率相关性分析 |
| 预期研究进度 | 4年 |

# 目录

| _, | 研究背景 | 7 |
|----|-----------------------------------|----|
| Ξ, | 研究目的 | 7 |
| 三、 | 研究对象 | 7 |
| | 3.1 纳入排除标准 | 7 |
| | 3.2 人工关节感染 MSIS 诊断标准(2014 版) | 8 |
| | 3.3 中止、终止临床研究的标准及剔除标准 | 8 |
| 四、 | 研究内容与方法 | 9 |
| | 4.1 收集受试者基线数据 | 10 |
| | 4.2 收集受试者术后抗生素使用情况 | 10 |
| | 4.3 监测受试者感染清除情况 | 10 |
| | 4.4 将受试者是否联合使用利福平与受试者感染清除情况进行对比分析 | 10 |
| 五、 | 临床试验实施方案 | 10 |
| | 5.1 研究周期 | 10 |
| | 5.2 具体研究流程 | 11 |
| | 5.3 随访要求 | 12 |
| | 5.4 研究流程图 | 13 |
| | 5.5 研究方案的调整或终止研究 | 13 |
| 六、 | 疗程前的检查 | 13 |
| | 6.1 筛选期及基线期的调查项目 | 13 |
| 七、 | 抗生素的使用方式、剂量、时间及疗程 | 14 |
| | 7.1 抗生素来源 | 14 |
| | 7.2 抗生素治疗的剂量、方式及疗程 | 14 |
| | 7.3 临床监护 | 14 |
| 八、 | 指标及评定标准 | 14 |
| | 8.1 主要疗效指标 | 14 |
| | 8.2 次要疗效指标 | 15 |
| 九、 | 安全性评价 | 15 |
| | 9.1 不良事件 | 15 |
| | 9.2 严重不良事件 | 15 |
| | 9.3 不良事件的记录与报告 | 15 |
| | 9.4 突发事件 | 16 |
| | 9.5 应急预案 | 16 |
| 十、 | 统计分析 | 17 |
| | 10.1 统计分析计划 | 17 |
| | 10.2 分析数据集 | 17 |
| | 10.3 缺失值的处理 | 17 |
| | 10.4 统计分析方法 | |
| | 10.5 统计软件与一般要求 | 19 |
| | 10.6 期中分析 | 19 |
| +- | 一、数据管理 | 19 |
| | 11.1 病例报告表的填写 | 19 |
| | 11.2 数据审核与分析 | 19 |

| 十二、 | 质量管理 | 19 |
|-----|-----------------|----|
| | 2.1 临床研究前培训 | |
| 12 | 2.2 提高受试者依从性的措施 | 20 |
| 十三、 | 质量控制和质量保证 | 20 |
| 十四、 | 伦理学要求和受试者知情同意书 | 20 |
| 十五、 | 资料保存 | 21 |
| 十六、 | 研究进度 | 21 |
| 十七、 | 附件 | 21 |

# 抗生素联合利福平治疗葡萄球菌假体周围感染的疗效与并 发症——一项多中心、随机对照试验

#### 一、研究背景

假体周围感染(Periprosthetic Joint Infection, PJI)是关节置换术后最具挑战性且严重的并发症之一。随着全球范围内关节置换手术的广泛开展,PJI 的发病率也随之上升,促使临床医生需要不断探索更有效的治疗方案。在 PJI 的治疗方案中,抗生素治疗尤为重要。PJI 的大部分致病菌为葡萄球菌,这些细菌都具有较强的生物膜形成能力,利福平,作为一种广谱抗生素,因其独特的抗菌机制和良好的组织穿透性,在 PJI 的治疗中扮演着不可或缺的角色,被广泛用于多种细菌感染特别是生物膜相关顽固性 PJI 的抗生素治疗中。

虽然目前多数研究表明抗生素联合利福平治疗能有效提高 PJI 的疗效,指南也推荐在葡萄球菌 PJI 外科手术治疗后,使用抗生素联合利福平治疗 3 个月,但既往文献证据并不充分,目前关于在葡萄球菌 PJI 抗生素治疗中是否添加利福平仍存在不同观点。既往关于利福平在 PJI 治疗中的应用相关研究大多为回顾性分析,因此可能存在选择偏倚、生存偏倚及其他混杂因素。目前仅有两项随机对照试验研究了利福平联合治疗在 PJI 中的效果,这些试验样本量都较小,且关于是否联合利福平治疗的结论并不一致。因此需要开展大规模的多中心随机对照试验,以明确利福平联合治疗是否有助于 PJI 感染的控制。

#### 二、研究目的

本研究拟设计一项多中心随机对照临床试验,旨在探讨利福平在葡萄球菌 PJI 抗生素治疗中临床价值。

#### 三、研究对象

选择在福建医科大学附属第一医院和其他分中心接受 DAIR 或移除假体翻修术且符合 入组标准的葡萄球菌 PJI 患者。

#### 3.1 纳入排除标准

#### 3.1.1 纳入标准

- ①根据 MSIS 标准确诊为 PJI
- ②经微生物培养确定致病菌为葡萄球菌并进行药敏测试
- ③有完整临床资料

- ④年龄<80周岁,没有严重的合并症或免疫抑制状态
- ⑤患者自愿参与本研究,并在身体与精神上可耐受本研究的治疗过程和各项检测,已签署知情同意书,并通过所有参与本研究的医院伦理委员会审核

#### 3.1.2 排除标准

- ①术前其他部位有慢性炎症者
- ②非葡萄球菌感染或混合感染者
- ③患者存在其他可能影响结果的疾病,如免疫缺陷、肝肾功能不全
- ④预期寿命小于半年者
- ⑤研究者判断患者因依从性问题不再符合该研究的标准
- ⑥对利福平过敏者

#### 3.2 人工关节感染 MSIS 诊断标准 (2014 版)

- 3.2.1 主要诊断指标(满足以下2条中任意1条):
  - 1) 存在与假体相通的窦道;
  - 2) 受累人工关节的 2 处假体周围组织或关节液标本中分离出同一病原体。
- 3.2.2 次要诊断指标(满足以下5条中任意3条):
  - 1) 红细胞沉降率 (ESR>30)或 C 反应蛋白 (CRP>10)水平升高;
  - 2) 关节液白细胞计数升高 (>3000)或白细胞酯酶试纸条测试结果 (++);
  - 3) 关节液中性粒细胞(PMN)百分比升高 (>80%);
- 4)阳性病理表现:400倍放大率下,假体周围组织的病理学分析在5个高倍镜视野下发现>5个中心粒细胞;
  - 5) 假体周围组织或关节液标本中1次培养分离出微生物。

## 3.3 中止、终止临床研究的标准及剔除标准

### 3.3.1 中止标准

- 1) 受试者根据自己意愿可随时退出研究;
- 2) 违反研究方案者且影响评估者;
- 3) 受试者发生不良事件且不能耐受者;

- 4) 研究者从医疗角度考虑不宜继续参加研究者。
- 5) 退出研究的受试者一定要问其退出的原因以及是否存在任何不良事件。需要时进行全面的评价,并尽可能做到详尽。如果可能,研究者也应该对这些受试者进行随访和评价。中止研究的原因必须记录。

#### 3.3.2 终止标准

- 1) 严重的治疗相关的不良事件;
- 2) 已经得出阳性的结论和有利的结果;
- 3) 在研究中发现临床研究方案有重大失误,难以评价治疗效应,或者一项设计较好的方案在实施中发生了重要偏差,再继续下去难以评价治疗效应;
  - 4) 课题负责单位要求终止(如经费原因、管理原因等)。

#### 3.3.3 剔除标准

- 1) 不符合入选标准者;
- 2) 符合排除标准者;
- 3) 无任何记录者:
- 4) 研究期间如加用其它治疗,经研究者评估影响研究评价者。

#### 四、研究内容与方法

本研究旨在评估 PJI 患者在外科治疗术后,联合使用利福平进行抗生素治疗在 PJI 中的疗效和安全性。研究对象为病原菌仅为葡萄球菌的 PJI 患者,按照严格的纳入和排除标准筛选入组,在接受 DAIR 或移除假体的翻修术后,随机分配至抗生素联合利福平治疗组或仅接受常规抗生素治疗组,然后对患者进行系统随访,定期评估其感染复发率、炎症指标、假体功能恢复及药物副作用等安全性指标。数据将通过统一的记录系统录入,并根据预定退出标准剔除不符合研究设计的患者。随访结束后,将数据汇总并进行分析,重点考察抗生素联合利福平治疗对 PJI 感染控制的有效性。通过该研究,我们希望明确利福平联合抗生素治疗在PJI 中的疗效和安全性,从而为 PJI 抗生素方案的优化提供参考依据。

DAIR 术后,结合既往回顾性分析结果,抗生素联合利福平治疗 PJI 感染控制率为 67.8%,单纯抗生素治疗 PJI 感染控制率为 45.78%,取  $\alpha$  值=0.05,  $\beta$  =0.9,抗生素联合利福平治疗组与抗生素治疗组样本比例为 1:1,失访率为 10% ,计算样本量:每组样本量需为 115 例,总共 230 例。

移除假体翻修术后,结合既往回顾性分析结果,抗生素联合利福平治疗 PJI 感染控制率为 85%,单纯抗生素治疗 PJI 感染控制率为 64.5%,取  $\alpha$  值=0.05, $\beta$ =0.9,抗生素联合利福

平治疗组与抗生素治疗组样本比例为 1:1,失访率为 10%,计算样本量每组样本量需为 89例,总共 198 例。

#### 4.1 收集受试者基线数据

收集受试者的基本信息、初次人工关节置换信息、DAIR 手术信息、翻修手术入院术前体格检查与辅助检查信息和 DAIR 手术信息、翻修手术信息作为基线数据,具体收集项目详见 CRF 表格。

#### 4.2 收集受试者术后抗生素使用情况

分别收集受试者抗生素使用情况,包括使用抗生素名称、单次剂量、频次、用药方式及 疗程等内容。

#### 4.3 监测受试者感染清除情况

在术后抗生素治疗开始后即开始监测受试者的感染清除情况,分别于手术后在抗生素治疗后 12 周、24 周、48 周、72 周和 96 周进行随访,随访方式包括返院复查和远程随访。

随访期间对受试者进行临床症状、体征的问诊与查体并记录;同时对患者进行实验室检查及影像学检查。根据 Claudio Diaz-Ledezma MD 等人提出的评估方法(附件六)判断患者的感染清除情况。

#### 4.4 将受试者是否联合使用利福平与受试者感染清除情况进行对比分析

首先,我们对受试者抗生素治疗方案和受试者感染清除情况进行描述性分析,明确受试者抗生素治疗方案,并计算受试者总体感染清除率;其次,根据受试者手术类型、抗生素方案及其他相关指标进行分层分析,控制混杂因素对研究结果的影响。最后,进行利福平联合抗生素治疗与感染清除率的相关性分析,评估抗生素联合利福平治疗组和单纯抗生素治疗组组间是否存在统计学差异,并进一步筛选影响感染清除疗效的相关因素。

#### 五、临床试验实施方案

#### 5.1 研究周期

## 5.1.1 受试者入组时间

患者签署《知情同意书》后,研究者根据入选排除标准对受试者进行筛选,筛选合格的 患者入组。

#### 5.1.2 研究持续时间

本试验在福建医科大学及其他合作中心等三甲医院中开展,基于各中心 PJI 患者的诊治

例数、各地区开展知情同意及各地区患者维持随访的难度,各中心竞争性入组,预计入组期为2年,考虑前期项目准备、随访复查、后期统计分析和临床试验总结报告审核等,本研究总体持续时间预计4年。

#### 5.1.3 受试者的预期参与时间

每位受试者预期参与持续时间约为2年,包含筛选入组期、基线期、治疗期以及随访期。

#### 5.2 具体研究流程

#### 5.2.1 临床研究 PI 筛选符合条件的受试者

#### 5.2.2 基线期临床资料收集

- 1) 基本信息:记录受试者出生日期、年龄、性别、民族、家庭住址及联系方式等资料
- 2) 体格检查:记录受试者的身高、体重、身体质量指数(BMI)、体温、血压、呼吸、脉搏等资料。
- 3) 症状体征:记录受试者 PJI 治疗前关节感染相关症状,包括发热、关节肿胀、关节周围皮温升高、切口红肿、窦道形成等资料。
  - 4) 功能评估: VAS 疼痛评分、KSS 膝关节功能评分、Harris 髋关节功能评分。
  - 5) 既往病史:疾病史和过敏史、疫区旅游史,年龄校正查尔森合并症指数。
- 6) 烟酒史:记录受试者的吸烟情况:日吸烟数量及吸烟年限;饮酒情况:如饮酒频率、 饮酒种类、饮酒数量、年限等。
- 7) 临床诊断:记录受试者入组时的临床诊断,如诊断名称、临床类型、病程(急性或慢性)等情况以了解受试者合并症情况。
- 8) 血常规检查(PJI治疗前):包括红、白细胞总数、血红蛋白(Hb)、血小板(PLT)、中性粒细胞计数(N)等。
- 9) 生化检查(PJI治疗前):包括谷丙转氨酶(ALT)、谷草转氨酶(AST)、总胆红素(TBIL)、总蛋白(TP)、白蛋白(ALB)、空腹血糖、糖化血红蛋白、肌酐、尿素氮、肾小球滤过率(GFR)、甘油三酯(TG)、胆固醇(TC)、低密度脂蛋白(LDL)、高密度脂蛋白(HDL)、钾、钠、氯、钙、磷等。
- 10) 凝血功能(PJI治疗前):包括凝血酶原时间(PT)、国际标准化比值(INR)、活化部分凝血活酶时间(APTT)、纤维蛋白原(Fib)、D-二聚体(D-dimer)
- 11) 炎症指标(PJI 治疗前):包括 C 反应蛋白(CRP)、红细胞沉降率(ESR)、降钙素原(PCT)、IL-6、D 二聚体、纤维蛋白原等。

- 12) 关节液检查(PJI治疗前):包括关节液白细胞计数、中性粒细胞比例以及关节液细菌培养等。
  - 13) 用于排除其他部位感染的实验室检查: 尿常规、粪常规、痰培养等
  - 14) 影像学检查(PJI治疗前):病变关节的 X线片、胸部 X线或 CT 检查
  - 15) 初次人工关节置换信息:记录受试者的置换部位、置换原因及感染部位等
- 16) 手术信息: 手术类型、手术时间、手术名称、手术时长、术中抗生素使用情况、关节液检查及细菌培养、组织病理检查等。
- 17) 抗生素使用情况:包括术后住院期间静脉使用抗生素及出院后抗生素治疗信息,具体收集抗生素名称、单次剂量、使用频率、使用方法、起止时间及使用天数等。

#### 5.2.3 随访

- 1) 随访方式: 返院复查、远程随访。
- 2) 随访时间:入组后均随访至少2年,分别于PJI 手术治疗后12周、24周、48周、72周和96周进行随访,随访方式包括返院复查和远程随访。
  - 3) 突发事件随访: 出现下述事件时,则立即进行一次随访
  - (1) 患者因感染再发再次入院治疗
  - (2) 患者因再植手术术后其他并发症再次入院治疗。

#### 5.2.4 观察终点

- 1) 假体周围感染再发:表现为出现感染的临床症状及体征或 CRP 指标上升,需要持续抗生素抑制治疗或手术治疗;
  - 2) 死亡;
  - 3) 随访时间超过24月,研究者判定为随访结束。
- 5.2.5 统计分析: 详见《十四、研究数据的统计分析》
- 5.2.6 向 IMCG 递交研究报告。
- 5.2.7 结题。

#### 5.3 随访要求

每次随访要求患者尽量到达手术医院进行,如无法到达需在当地医院进行相应检查,并电话随访。研究者需对患者的感染状态进行评估,感染状态评估的参考指标包括但不限于: 发热、局部皮温升高、关节肿胀、切口红肿、窦道、红细胞沉降率 (ESR>30)或 C 反应蛋白 (CRP>10)水平升高。

每次随访需进行相应的检查项目,包括生命体征、体格检查、疼痛评分、功能评分、血

常规、CRP、ESR、生化、凝血功能、尿常规及影像学检查等,具体随访要求参考研究流程表 (附件七)。

#### 5.4 研究流程图



图 1: 本研究的研究流程图

### 5.5 研究方案的调整或终止研究

鉴于本研究的相关临床研究已经在国内外多家大型医院完成了至少超过 300 例的临床 治疗,证实其结果是安全和可靠的,并且本研究不对临床抗生素用药方案进行干预,仅记录 用药后的疗效。因此,我们有理由相信本研究能够顺利实施。如果研究方案有重大调整和修 改或需要终止,需在上述确定性的临床结果基础上由专家委员会共同讨论后决定及实施。

#### 六、疗程前的检查

#### 6.1 筛选期及基线期的调查项目

- 1) 术前完整的病史采集、体格检查(包括切口情况、局部皮温、压痛、有无窦道、VAS 疼痛评分、关节功能评分(髋关节: Harris 膝关节: KSS)) 及生命体征的记录;
- 2) 术前实验室检查项目: 血常规、尿常规、便常规+潜血,生化全项(包括 ALT、AST、LDH、GGT、ALP、CK、CKMB、TBIL、IBIL、BUN、Cr、UA、ALB、Ca<sup>2+</sup>、Mg<sup>2+</sup>、P<sup>3+</sup>、K<sup>+</sup>、Na<sup>+</sup>、CL<sup>-</sup>、GLU、INR、APTT、PT、D-dimer、SCRP、BNP)血清炎症指标(CRP、ESR),以及 PJI 保留假体或翻修手术术中检查结果(包括关节液白细胞计数和分类,术中冰冻结果,术中培养结果);

- 3) 术前辅助检查项目(包括患侧关节正侧位片,胸部平片或CT,根据个人情况的其他 检查):
  - 4) 从既往病历中搜集可获得的初次关节置换的信息。

#### 七、抗生素的使用方式、剂量、时间及疗程

#### 7.1 抗生素来源

本研究所使用常规抗生素治疗,作为基础治疗方案,由患者自负费用。利福平治疗,作为研究干预措施的一部分,若患者被分配至利福平联合抗生素治疗组,将在常规抗生素治疗基础之上,额外口服利福平三个月。利福平的市场单价为 22.93 元人民币,药品规格为 0.15 克×100 粒。作为本研究的一部分,在研究期间使用利福平的费用不由患者承担。

#### 7.2 抗生素治疗的剂量、方式及疗程

在葡萄球菌 PJI 抗生素的选择中,将根据病原菌的药敏结果选择相应的抗生素治疗:

- 1) 静脉:针对甲氧西林敏感的葡萄球菌,选择头孢唑林进行静脉抗生素治疗;针对耐甲氧西林的葡萄球菌,选择万古霉素进行静脉抗生素治疗。静脉抗生素治疗周期为 2-3 周;
- 2) 口服:静脉抗生素治疗结束后,改为口服进行抗生素治疗:如果葡萄球菌对氟喹诺酮类抗生素敏感,则选择氟喹诺酮类口服进行治疗;如果葡萄球菌对氟喹诺酮类抗生素耐药,则选择利奈唑胺口服进行治疗。根据说明书进行抗生素治疗。抗生素联合治疗组还另外联合使用利福平,利福平给药方案:10mg/kg,总剂量在0.6-0.9g/天。口服抗生素治疗周期为3个月。

#### 7.3 临床监护

对于所有受试者,住院期间每天均对受试者进行评估,出院期间前按研究要求时间点进行评估。对于完成治疗后进入随访期的受试者,应至少每3个月进行一次随访。

#### 八、指标及评定标准

#### 8.1 主要疗效指标

- 1) 感染的清除率,感染清除率计算公式:判定为感染清除的受试者例数/完成随访的受试者总例数。感染清除定义为患者(1) 感染根除,伤口愈合,无瘘管、无引流、无痛感,无同一菌种感染复发;(2) 无因感染再次手术干预;(3) 没有发生 PJI 相关疾病如败血症、坏死性筋膜炎等导致的死亡(详见附件六)。
  - 2. 与 PJI 相关的不良事件。

#### 8.2 次要疗效指标

- 1) 术后的功能评分;
- 2) 术后假体松动的比率、翻修率、需要移除假体所占比率;
- 3) 抗生素并发症的发生率。

#### 九、安全性评价

#### 9.1 不良事件

不良事件指治疗过程中或治疗后发生的不可预见的医疗状况,或者使原有医疗状况恶化的事件,其发生与所用治疗方案不一定有因果关系。不良医疗状况包括症状、体征和异常检查结果。在临床研究中,不良事件可以包括任何时间所发生的任何不可预见的不适。

#### 9.2 严重不良事件

严重不良事件是指在研究阶段(包括筛选期、治疗期和随访期)使用任何剂量的研究药物(包括对照药和安慰剂)导致的符合以下一项或多项标准的不良事件:

- (1) 致死
- (2) 危及生命
- (3) 需住院治疗或延长住院时间
- (4) 伤残、影响工作能力
- (5) 先天畸形
- (6) 致癌
- (7) 有重要的医学意义,需要医学处理来防止永久性的损伤或损害(指不会立即危及生命或导致死亡或住院的事件,但可能危害受试者或需要采取措施来预防上述所列情况发生的医疗事件,如:如血管神经性水肿,暂不需要气管插管但需要皮质激素治疗的事件;需要强化治疗的过敏性支气管痉挛等)

#### 9.3 不良事件的记录与报告

应当在整个研究过程中注意不良事件的收集和记录。

- 9.3.1 不良事件应记录的内容如下:
  - (1) 不良事件的描述
  - (2) 发生和停止时间
  - (3) 程度及发作频度
  - (4) 采取的相应措施

- (5) 与治疗的因果关系
- (6) 转归
- (7) 判断是否为严重不良事件。

有关不良事件的医学文件应记录在原始病历中,包括实验室检查的通知单(如: x 线检查、心电图等)和检查结果报告单。如受试者因研究结束或受试者出院等而无法继续接受研究者的治疗,研究者应将受试者的病历摘要(包括治疗安排和不良事件是否需要继续随访的说明等)交给负责继续治疗的研究者。这些信息也要记录在原始病历中。突发事件是临床研究中突然发生,造成或可能造成受试者损害,需要医护人员紧急处理的事件

#### 9.3.2 严重不良事件的记录与报告

在研究过程中发现任何严重不良事件,研究者或中心相关人员都必须在获知后的 24 小时内通报给主要研究者、伦理委员会和课题负责单位。课题负责单位将协助研究者以获得严重不良事件所必须的信息,并确保课题负责单位在规定的时间内获得相应的报告,并在规定时间内上报当地监管部门。同时研究者必须填写严重不良事件表,记录严重不良事件的发生时间、严重程度、持续时间、采取的措施及转归等。

如非严重不良事件进展为严重不良事件,该事件及相关报告也必须在获知后的 24 小时内通报。

| 单 位 | 联系人 | 电话 | 传真 |
|--------------------|-----|---------------|---------------|
| 福建医科大学附属第一医院 伦理委员会 | 刘媛 | 0591-87981029 | 0591-87981028 |

#### 9.4 突发事件

突发事件是临床研究中突然发生,造成或可能造成受试者损害,需要医护人员紧急处理 的事件

#### 9.5 应急预案

- (1) 预防为主:发现病例,及时报告,积极采取有效措施控制病情发展。
- (2) 依法管理:在临床试验中,贯彻执行相关法律法规,对突发事件和不良事件及时报告,在整个控制和救治过程中实行已发管理。
- (3)分级负责:在临床试验中,充分发挥"三级质量监控"(申办方监察员、专业科室、机构办公室),严格执行标准化操作规程,定期或不定期检查、督查整个过程,做到即时发现,即时救治。
  - (4) 快速反应: 建立预警和医疗救治快速反应,强化人力、物力、财力储备,增强应

急处理能力,按照早期发现,及时报告,依靠科学,措施果断的原则,及时准确处理。

### 十、统计分析

#### 10.1 统计分析计划

统计分析计划将在研究开始后开始制定,并于数据库锁定前确定。计划内需包含所有统计学分析将要涉及的内容,包括用于分析的数据集的定义和不同指标采用的统计学描述和分析方法等。

由于方案的更改导致原定统计分析计划的变动,应与申办方、研究者、数据管理和统计分析方以及伦理等多方之间达成共识,并严格遵守临床试验操作规章流程进行改动,否则不宜轻易进行更改。

#### 10.2 分析数据集

10.2.1 全分析集(FAS):指合格病例和脱落病例的集合,但不包括剔除病例。对基线分析和人口学特征等作可比性分析。主要疗效指标缺失时,根据意向性分析(intention to treat,ITT 分析)原则,用前一次结果结转。可比性分析和次要疗效指标的缺失值不作结转(data-carry-forward),根据 FAS 中实际获得的数据分析。

10.2.2 符合方案集(PPS): 指符合纳入标准、不符合排除标准、完成治疗方案的病例集合,即对符合研究方案、依从性好、完成 CRF 规定填写内容的病例进行分析(PP 分析)。PP 分析主要用于主要疗效指标。

10.2.3. 安全数据集(SS): 至少接受一次治疗,且有安全性指标记录的实际数据。安全性缺失值不得结转;纳入可作评价的部分剔除病例,如年龄超过纳入标准的病例,但不包括使用禁用药物导致无法作安全性判断的病例。不良反应的发生率以安全集的病例数作为分母。

#### 10.3 缺失值的处理

对于研究过程中可能出现的缺失数据,分析时仅针对主要终点指标的缺失进行结转。采用单值结转的方法,通过 LOCF(Last Observation Carry Forward)策略对主要终点的缺失数据进行结转。对于其他指标的缺失,将不进行结转处理。

错误及不合理数据将在统计分析之前的数据清理过程予以处理。对于中途退出或撤出试验,此部分患者信息仍将被纳入最终的统计分析。统计报告中,将对所有退出或撤出患者的具体原因进行详细说明,有与早期退出导致的主要指标缺失,将按照上述的缺失值处理策略

进行结转。

#### 10.4 统计分析方法

#### 10.4.1 一般原则

所有的统计检验均采用双侧检验,p值<0.05 将被认为所检验的差别有统计学意义(特别说明的除外)。计量资料的描述将计算均值、标准差、中位数、最小值、最大值、下四分位数(Q1)和上四分位数(Q3),计数资料采用例数及百分数表示。本组研究主要针对是否联用利福平治疗对 PJI 感染再发的影响,故组间比较将根据 5 年内感染再发对的分布情况采用卡方检验或精确概率法(若卡方检验不适用)。

#### 10.4.2 完成情况及受试者分布

总结各中心及整体筛选、入组及完成病例数、各分析集病例分布情况,对脱落原因和未进入 FAS 原因分别进行分类汇总,并列出脱落及未进入 FAS 的受试者清单。分别描述各中心病例入组及完成情况,总结相应统计分析人群的情况,列出不符合试验方案入选、病例剔除、病例脱落详细情况。各组不同数据集大小、各中心病例分布、总脱落率比较、未完成原因详细列表。

#### 10.4.3 受试者基线数据分析

基线数据分析在 FAS 中进行。基线数据定义为受试者 PJI 手术治疗前的最后一次非缺失的数据。针对病例入组时人口学特征、相关检查、检测指标等,以观察各组基础情况是否可比。其中,定量指标列出例数、均数、标准差、中位数、最大值、最小值;定性指标,列出频数及百分数。基线资料均衡性分析:对人口学等资料、一般情况及临床情况进行描述。

#### 10.4.4 受试者随访期数据分析

分别描述受试者术后抗生素方案及感染清除率。计量数据用Shapiro-Wilk法进行正态性检验,若数据符合正态分布,则结果用均数土标准差表示,并计算其95%置信区间(95% CI),若不符合正态分布,数据用下四分位数(Q1)和上四分位数(Q3)表示。受试者总体感染清除率计算公式为:判定为感染清除的受试者例数/完成随访的受试者总例数。感染清除定义为患者无感染的临床症状、体征,直至随访终点没有因感染复发而再次手术或需要长期抗生素抑制治疗。

## 10.4.5 分层分析与倾向性分层分析

1)分层分析:将手术方式作为分层变量,以每种手术的单纯抗生素治疗组作为参照组, 比较不同手术方式是否影响联用利福平对 PJI 的治疗效果。 2)倾向性分层分析:根据分组,对比各组患者的基线资料特征,将混杂因素如受试者年龄、性别、感染部位、感染病原体、糖尿病、手术方式等纳入倾向性分析,构建 Logistic回归模型,其中因变量为是是否联合利福平治疗,自变量为混杂因素,计算倾向性评分。将倾向性评分进行五分位分层,再分析是否联合利福平治疗与关节感染再发的关系。

#### 10.4.6 研究数据的相关性分析

主要评价指标(感染控制率)采用 Mantel-Haenszel 卡方检验联合 Cramer's V 检验进行相关性分析。根据分层分析的结果,将手术方式分组,因变量为各组受试者感染控制率,卡方检验分析 PJI 术后利福平治疗与受试者感染控制率的相关性统计学意义,Cramer's V 检验判断二者间的关联强度。

#### 10.5 统计软件与一般要求

采用 SPSS 20.0 软件分析。

所有的统计检验均采用双侧检验,P值小于或等于0.05将被认为所检验的差别有统计 意义。主要疗效指标将采用优效性检验,其他内容的统计分析将采用差异性检验。

详细的统计分析方法将在统计分析计划中提供。

#### 10.6 期中分析

设定在项目启动一年后进行期中分析,根据已收集的资料统计项目完成情况及受试者分布,进行受试者基线数据分析、受试者随访期数据分析、分层分析与倾向性分层分析。

#### 十一、数据管理

#### 11.1 病例报告表的填写

本研究的数据管理采用填写电子病例报告表(eCRF),原始记录、所有实验室检查结果应完整保存。研究中的任何观察、检查结果均应及时、准确、完整、规范、真实地记录于eCRF中,研究结束后交由课题负责单位进行统计分析。

#### 11.2 数据审核与分析

数据收集齐全后由研究者、统计分析人员对数据进行数据审核。数据审核后交统计人员 进行分析,同时定稿统计计划书,并按统计分析计划进行统计分析。

#### 十二、质量管理

研究的质控根据 ICH-GCP 进行。

#### 12.1 临床研究前培训

课题负责单位负责组织专家在临床研究开始前对研究者进行研究方案的培训,对症状体 征量化标准进行一致性测评。签署研究者声明。

课题负责单位及研究者均应履行各自职责,并严格遵循临床研究方案,采用标准操作规程,以保证临床研究的质量控制和质量保证系统的实施。

#### 12.2 提高受试者依从性的措施

研究者应认真执行知情同意,使受试者充分理解研究要求的基础上,完全自愿参与研究。

### 十三、质量控制和质量保证

为保证多中心研究的质量,在正式研究开始前,由参加研究的主要负责人,共同讨论、制定临床研究方案。对参加研究的有关医务人员进行同期培训。

临床研究中所有观察到的结果和异常发现,均应及时加以认真核实、记录,保证数据的可靠性。临床研究中各种检查项目所使用的各种仪器、设备、试剂、标准品等,均应有严格的质量标准,并确保是在正常状态下工作。临床数据的记录和转移,必须由有经验的医师负责,并有专人监督或核对,以保证数据的科学性和准确性。临床研究的各种结论,必须来源于原始数据。

研究者应完整、详细、准确、及时地填写病例报告表(CRF)。交主要研究者签名确认 后按规定程序报送或保存。所有与研究有关的数据资料应集中管理与分析。

建立数据保管、数据传递、数据查询的程序。保管的资料包括:受试者的原始病历、影像学资料、CRF、受试者筛选表、受试者鉴认代码表、严重不良事件报告表、访视报告表及有关的各种原始医疗文件等。传递的数据包括:受试者总随机表、CRF、严重不良事件报告表及总结资料需使用的数据和资料。

总结和分析临床研究结果时,必须采用规范的统计学分析方法,并请熟悉生物统计学的 人员参与。

#### 十四、伦理学要求和受试者知情同意书

本临床研究必须遵循《赫尔辛基宣言》中的伦理原则和国际有关药物临床研究的管理规范与法规。本研究开始前需报送资料(研究方案、病例报告表、知情同意书等)经单位伦理委员会审核,获得批准后方可开始研究。研究过程中如果确需对研究方案、CRF、知情同意书进行修改,须报单位伦理委员会审核批准后方可实施。

每一位受试者入选本研究前,研究者有责任向其和(或)法定代理人客观、全面地介绍本研究的目的、程序和可能的获益与风险。应让受试者知道他们有权决定是否参加本研究,

并有权要求中途不需要任何理由退出本研究。研究医师必须在每位受试者进入研究之前获得 受试者和(或)其法定代理人签署的知情同意书,并作为研究档案保存。

受试者出现不良事件应及时给予处理措施,直至不良事件消失或纠正到临床允许的状况。实验室异常指标要定期复查测定,直至临床允许的范围内为止。

出现严重不良事件,要积极抢救,并按照当地法规要求上报当地药监部门、研究单位伦 理委员会,并通知课题负责单位及其伦理委员会。

## 十五、资料保存

研究者必须保存每位受试者的原始资料(通常在受试者病历中),出现在 CRF 上的信息都应可以在这些原始资料中找到出处,原始资料包括:原始记录、受试者签署的知情同意书、实验室数据、影像学资料、心电图、用药记录等。

应按照规定对受试者的基本资料保存足够长时间(通常为研究结束后 5 年),基本资料包括:

- 1. 伦理委员会对研究方案及所有方案修订的批件;
- 2. 所有原始医疗文件:
- 3. 电子病历系统;
- 4. 己签署的知情同意书;
- 5. 其它研究相关文件。

#### 十六、研究进度

入组计划:本研究计划于2024年12月启动,预计入组时间从:2024-12至2025-12月。每2-3月召开工作组会议。第一年拟入组200例,第二年入组另外300例,以后的2年序贯治疗、观察疗效及安全性等。

### 十七、附件

附件一:人工关节感染MSIS诊断标准(2014版)

附件二: 关节疼痛VAS评分

附件三: 年龄校正查尔斯合并症指数

附件四: 髋关节功能Harris评分

附件五:膝关节功能KSS评分

附件六: 感染清除评估标准表

附件七: 研究流程表

附件八:知情同意书

附件九: 利福平的毒副作用及风险预案

#### 十八、参考文献

- [1] Rajput V, Meek RMD, Haddad FS. Periprosthetic joint infection: what next? Bone Joint J 2022;104-B:1193-5.
- [2] Kurapatti M, Oakley C, Singh V, Aggarwal VK. Antibiotic Therapy in 2-Stage Revision for Periprosthetic Joint Infection: A Systematic Review. JBJS Rev 2022;10.
- [3] Fisher C, Patel R. Rifampin, Rifapentine, and Rifabutin Are Active against Intracellular Periprosthetic Joint Infection-Associated Staphylococcus epidermidis. Antimicrob Agents Chemother 2021;65.
- [4] El Helou OC, Berbari EF, Lahr BD, Eckel-Passow JE, Razonable RR, Sia IG, Virk A, Walker RC, Steckelberg JM, Wilson WR, Hanssen AD, Osmon DR. Efficacy and safety of rifampin containing regimen for staphylococcal prosthetic joint infections treated with debridement and retention. Eur J Clin Microbiol Infect Dis 2010;29:961–7.
- [5] Zimmerli W, Sendi P. Role of rifampin against staphylococcal biofilm infections in vitro, in animal models, and in orthopedic-device-related infections. Antimicrob Agents Chemother 2019;63:1–10.
- [6] Beldman M, Löwik C, Soriano A, Albiach L, Zijlstra WP, Knobben BAS, Jutte P, Sousa R, Carvalho A, Goswami K, Parvizi J, Belden KA, Wouthuyzen-Bakker M, Wouthuyzen-Bakker M. If, when, and how to use rifampin in acute staphylococcal periprosthetic joint infections, a multicentre observational study. Clin Infect Dis 2021;73:1634–41.
- [7] Cortés-Penfield NW, Hewlett AL, Kalil AC. Adjunctive Rifampin Following Debridement and Implant Retention for Staphylococcal Prosthetic Joint Infection: Is it Effective if not Combined With a Fluoroquinolone? Open Forum Infect Dis 2022;9:1–4.
- [8] Zimmerli W, Widmer AF, Blatter M, Frei R, Ochsner PE. Role of rifampin for treatment of orthopedic implant-related staphylococcal infections: a randomized controlled trial. Foreign-Body Infection (FBI) Study Group. JAMA 1998;279:1537–41.
- [9] Leijtens B, Elbers JBW, Sturm PD, Kullberg BJ, Schreurs BW. Clindamycin-rifampin combination therapy for staphylococcal periprosthetic joint infections: A retrospective observational study. BMC Infect Dis 2017;17:1–7.
- [10] Scheper H, Gerritsen LM, Pijls BG, Van Asten SA, Visser LG, De Boer MGJ. Outcome of Debridement, Antibiotics, and Implant Retention for Staphylococcal Hip and Knee Prosthetic

Joint Infections, Focused on Rifampicin Use: A Systematic Review and Meta-Analysis. Open Forum Infect Dis 2021;8:ofab298.

- [11] Lora-Tamayo J, Murillo O, Iribarren JA, Soriano A, Sánchez-Somolinos M, Baraia-Etxaburu JM, et al. A large multicenter study of methicillin-susceptible and methicillin-resistant Staphylococcus aureus prosthetic joint infections managed with implant retention. Clin Infect Dis 2013;56:182–94.
- [12] Karlsen ØE, Borgen P, Bragnes B, Figved W, Grøgaard B, Rydinge J, Sandberg L, Snorrason F, Wangen H, Witsøe E, Westberg M. Rifampin combination therapy in staphylococcal prosthetic joint infections: a randomized controlled trial 2020;2:1–9.
- [13] Renz N, Trampuz A, Zimmerli W. Controversy about the Role of Rifampin in Biofilm Infections: Is It Justified? Antibiot (Basel, Switzerland) 2021;10.
- [14] Kusejko K, Auñón Á, Jost B, Natividad B, Strahm C, Thurnheer C, et al. The Impact of Surgical Strategy and Rifampin on Treatment Outcome in Cutibacterium Periprosthetic Joint Infections. Clin Infect Dis 2021;72:E1064–73.
- [15] Aydın O, Ergen P, Ozturan B, Ozkan K, Arslan F, Vahaboglu H. Rifampin-accompanied antibiotic regimens in the treatment of prosthetic joint infections: a frequentist and Bayesian meta-analysis of current evidence. Eur J Clin Microbiol Infect Dis 2021;40:665–71.
- [16] Gómez J, Canovas E, Baños V, Martínez L, García E, Hernández-Torres A, Canteras M, Ruiz J, Medina M, Martínez P, Canovas A, Soriano A, Clavel M. Linezolid plus rifampin as a salvage therapy in prosthetic joint infections treated without removing the implant. Antimicrob Agents Chemother 2011;55:4308–10.
- [17] Eriksson HK, Lazarinis S, Järhult JD, Hailer NP. Early Staphylococcal Periprosthetic Joint Infection (PJI) Treated with Debridement, Antibiotics, and Implant Retention (DAIR): Inferior Outcomes in Patients with Staphylococci Resistant to Rifampicin. Antibiotics 2023;12.

# 附件一: 人工关节感染 MSIS 诊断标准(2014版)

## 主要诊断指标 (满足以下 2条中任意 1条):

- 1) 存在与假体相通的窦道;
- 2) 受累人工关节的 2 处假体周围组织或关节液标本中分离出同一病原体。

### 次要诊断指标(满足以下5条中任意3条):

## 诊断指标

- 1) 红细胞沉降率 (ESR>30)或 C 反应蛋白 (CRP>10)水平升高;
- 2) 关节液白细胞计数升高 (>3000)或白细胞酯酶试纸条测试结果 (++);
- 3) 关节液中性粒细胞(PMN)百分比升高 (>80%);
- 4)阳性病理表现:400倍放大率下,假体周围组织的病理学分析在5个高倍镜视野下发现>5个中心粒细胞;
- 5) 假体周围组织或关节液标本中1次培养分离出微生物。

# 附件二: 关节疼痛 VAS 评分

视觉模拟评分(VAS)标准(0分-10分)

0分: 无痛;

3 分以下: 有轻微的疼痛, 能忍受;

4分-6分:疼痛影响睡眠,尚能忍受;

7分-10分:有较强烈的疼痛,疼痛难忍,影响食欲,影响睡眠

## 附件三:年龄校正查尔森合并症指数 (aCCI)

以下项目计1分

心肌梗死

充血性心衰

周围性血管病变

脑血管疾病

痴呆症

慢性阻塞性肺病

结缔组织病

消化性溃疡病

轻微的肝脏疾病

糖尿病

以下项目计2分

偏瘫

中/重度肾病

糖尿病办器官损害

任何肿瘤

白血病

淋巴瘤

以下项目计3分

中/重度肝病

以下项目计6分

转移性实体瘤

艾滋病

年龄

超过 40 岁每 10 岁分计 1 分; 即>50 计 0 分以上项目累加即为年龄校正查尔斯合并症指数。

# 附件四: 髋关节功能 Harris 评分

## Harris 髋关节评分表

姓名: 住院号: 部位: 左/右髋 联系电话: 评分日期: 编号:

| 火土 イ | | 上院与: 市位: 左/右腕 | <b>绷 勺:</b> |
|-----------|-----|----------------------------|-------------|
| | 疼 | 痛 (44) | |
| 无 | 无疼症 | Ħ | 44 |
| 轻 | 偶而纲 | 疼痛或者意识不到的轻微疼痛,不影响活动 | 40 |
| 微 | 不影响 | 向活动,加剧活动后很少引起中等程度的疼痛,可能服用阿 | 司匹 30 |
| | 林 | | |
| 中 | | T忍受,活动受到一些限制,但仍能正常工作,可能偶尔需 | 要服 20 |
| <u>'</u> | | 可司匹林药效更强的止痛药物 | |
| 著 | 经常发 | 文生严重疼痛,但能走动,活动严重受限,需要经常服用比 | 阿司 10 |
| 1 | 匹林刻 | <b>5效更强的止痛药物</b> | |
| 重 | 因严重 | <b>重疼痛而致残,卧床不起</b> | 0 |
| | | 功 能 (47) | |
| | | 不需借助扶手 4 | 4 |
| | 上 | 需借助扶手 2 | 2 |
| 日 | 楼 | 其他方式上楼 | 1 |
| | | 不能上楼 ( | 0 |
| 常 | 转移 | 可以乘坐公共交通工具 | 1 |
| | | 可以舒适地在任何高度的椅子上坐立1小时以上 : | 5 |
| 活 | 坐 | 可以舒适地在高位椅子上坐立半小时以上 | 3 |
| <b>→1</b> | | 不能在任何高度的椅子上坐立 ( | 0 |
| 动 | 穿 | 可轻松完成 4 | 4 |
| | 鞋 | 有困难但能完成 2 | 2 |
| | 袜 | 不能完成 | 0 |
| | | 无 [ | 11 |
| | 跛 | 轻度 8 | 8 |
| | 行 | 中度 | 5 |
| | | 重 | 0 |
| 步 | | 不需要 | 11 |
| | 行 | 长途行走时需要手杖 | 7 |
| | 走 | 大多数行走时需手杖 : | 5 |
| | 支 | 需单拐 3 | 3 |
| | 持 | 双手杖 2 | 2 |
| 态 | | 双拐 | 0 0 |

| | | 不能 | <b></b><br>能行走 | | 0 | |
|---|---|---|---|---|---|---|
| | 行 | 无肾 | 艮制 | | 11 | |
| | 走 | 6 | 个街区, | 约 600m | 8 | |
| | 距 | 2-3 | 街区, | 约 200-300m | 5 | |
| | 离 | 只負 | <b></b> | 7活动 | 2 | |
| | | 只負 | <b></b> 能在床上 | _活动 | 0 | |
| | Γ | | | 关节活动度 (5) | | |
| | 0-45° | | ( ) | ×1.0×0.05 | | |
| | 46-90° | | {[( | )-45°]×0.6+45}×0.05 | | |
| 屈 | 91-110 | )° | {[( | )-90°]×0.3+72} ×0.05 | | |
| | ≥111° | | 3.9 | | | |
| 伸 | 任何 | 角 | 0 | | 0 | |
| -14 | 度 | | ( ) | 0.0.005 | | |
| 外屋 | 0-15° | | | ×0.8×0.05 | - | |
| 展 | 16-20° | | {[( | )-15°]×0.3+12]}×0.05 | - | |
| | 21-45 | | 0.675 | 0.0.0.5 | | |
| 内 | 0-15° | | , , | ×0.2×0.05 | - | |
| 收<br>外 | ≥16°<br>0-15° | | 0.15 | V0 4V0 05 | | |
| 旋 | 0-15°<br>≥16° | | 0.3 | ×0.4×0.05 | | |
| 内 | 任 何 | - 白 | 0.3 | | 0 | |
| 旋 | 度 | 川 | U | | 0 | |
| 74/- | | | | 肢 体 畸 形 (4) | | |
| 屈曲 | 事缩< | 30° | | 100 11 1 10 10 | 1 | |
| | 了。<br>【畸形< | | | | 1 | |
| | | 1 | | | | |
| 肢体 | 本不等长 | <3 | .2cm | | 1 | |
| | | | | | 总 | 分: |
| exce | ellent ( | => 9 | 0) go | ood (80-89) fair (70-79) poor (< 70 | ) 评 | : |
| 价等 | 穿级: | | | | | |
| | | | | 31 3 - 13 - 13 - 13 - 13 - 13 - 13 | | |

注: 内外旋检查时应为髋伸直位

## 附件五: 膝关节功能 KSS 评分

## 膝关节功能评分表(KSS)

 姓名:
 住院号:
 临床诊断:
 术式:

 第 次
 记录时间:
 年 月 日

第\_\_\_\_次 总分

疼痛评分(如总分为负数,得分为0) 疼痛 不疼 50 偶尔觉轻微疼痛 45 上楼时偶尔轻微疼痛 40 上楼和走路时偶尔轻微疼痛 30 中度疼痛 偶尔疼得比较厉害 20 经常疼得比较厉害 10 疼得特别厉害,需要服药 0 活动度 由屈曲到伸膝 每5°得1分 稳定性(在任何位置 前后侧 <5mm 10 上的最大活动度) (10)5~10mm 5 0 >10mm 内外侧 <5° 15 (15) 6°∼9° 10 10°∼14° 5 0 >15° -2 减分 屈曲挛 5°~10° 缩(-15) 10°~15° -5 -50  $16^{\circ}{\sim}20^{\circ}$ -10 -15 >20° 伸展缺 <10° -5 损(-15) 0°~20° -10 >20° -15 对 线 | 外翻 5°~10° 0分 (-15) 内翻 0°~4° 每度减3分 每度减3分 外翻 11°~15° 其他 -20分 功能评分(总评分为各项之和) 行走能力 50分 无任何限制 50

抗生素联合利福平治疗葡萄球菌假体周围感染的疗效与并发症———项多中心、随机对照试验 版本号 V2.0 福建医科大学附属第一医院 版本日期: 2024 年 10 月 12 日

| | | 约1公里以上 | 40 |
|-----|-----|-------------------|-----|
| | | 500-1000 米 | 30 |
| | | 不到 500 米 | 20 |
| | | 仅能在室内活动 | 10 |
| | | 不能步行 | 0 |
| 上下楼 | | 正常上下楼梯 | 50 |
| | | 正常上楼梯,下楼梯借助扶手 | 40 |
| | | 需借助扶手才能上下楼梯 | 30 |
| | | 借助扶手能上楼梯,但不能独立下楼梯 | 15 |
| | | 完全不能上下楼梯 | 0 |
| 减分 | -20 | 用手杖 | -5 |
| | | 用双手杖 | -10 |
| | | 需使用腋杖或助行架辅助活动 | -20 |

附注 1: 85~100 分 优 ; 70~84 分 良 60~69 分 可 ; <60 分 差

附注 2: 方框内标有"分"的填具体分数;

方框内标有""的填具体度数;

方框内无任何标志的只需在相应项打"√",肌力项除外。

# 附件六:感染清除评估标准表

| | 无临床症状(伤口愈合,无瘘管或引流,关节无痛); |
|----------------------|-------------------------------|
| | 血清学标志物(包括 C 反应蛋白、红细胞沉降率、白细 |
| | 胞)恢复到基线(或正常水平); |
| A. 感染根除: | 无需抗生素抑制治疗; |
| | 无由同一生物菌株引起的感染复发; |
| | 没有发生(新的)不同微生物的感染; |
| | 在其他手术部位没有伴随的 PJI。 |
| | 未因感染再次手术; |
| | 在随访期内未因无菌性原因进行翻修(包括无菌性松 |
| B.手术后无因感染再次手术干预: | 动、不稳定、僵硬); |
| | 再植入术后未进行其他手术治疗(包括:下肢截肢、髋 |
| | /膝关节固定术、髋关节切除术)。 |
| | 无因与 PJI 直接相关的疾病(包括败血症、坏死性筋膜 |
| | 炎)导致死亡; |
| | 无因 PJI 治疗住院死亡,原因与 PJI 无直接关联(包 |
| C 不去去 DII 机光式运用水物压力 | 括心肌梗死、中风、肺炎); |
| C.不存在 PJI 相关疾病导致的死亡: | PJI 治疗期间住院时间少于 3 个月/年; |
| | 无与 PJI 静脉或局部抗生素治疗相关的医疗并发症 |
| | (包括全身毒性、肾功能不全、外周插入中央导管并发 |
| | 症)。 |

表格引用自: Diaz-Ledezma C, Higuera CA, Parvizi J. Success After Treatment of Periprosthetic Joint Infection: A Delphi-based International Multidisciplinary Consensus[J]. Clinical Orthopaedics and Related Research®, 2013.

# 附件七: 研究流程表

| | 筛选 | | 治疗 | | <br>抗 <u></u> | 生素治疗 | <br>后随访其 | <br>玥 | |
|---|---|---|---|---|---|---|---|---|---|
| 调查项目 | 期 | 基线期 | 期 | V1 | V2 | V3 | V4 | V5 | V6 |
| 签署知情 | | | | | | | | | |
| 同意书 | × | | | | | | | | |
| 入排标准 | × | | | | | | | | |
| 基本资料 | | × | | | | | | | |
| 体格检查 | | × | × | × | × | × | × | × | × |
| 症状体征 | | × | × | × | × | × | × | × | × |
| 既往史 | | × | | | | | | | |
| 血常规 | | × | × | × | × | | × | | × |
| 炎症指标 | | × | × | × | × | | × | | × |
| 关节液检 | | | | | | | | | |
| 查 | | × | | | | | | | |
| 组织病理 | | × | | | | | | | |
| 血生化 | | × | × | × | | | | | |
| 凝血功能 | | × | | | | | | | |
| 尿常规 | | × | | | | | | | |
| 患侧关节 | | | | | | | | | |
| X线 | | × | × | × | × | | × | | × |
| 抗生素并 | | V | | | \ | | V | | |
| 发症 | | × | × | × | × | | × | | × |
| 手术相关 | | | | | | | V | | |
| 并发症 | | | | × | × | | × | | × |
| 感染状态 | | × | | × | × | | × | | × |

| 评估 |
|----|

#### 注:

- 1、筛选期为PJI治疗手术入院时。×:必须收集的信息,余为可选收集信息。
- 2、基线期为PJI治疗手术入院检查以及既往病史的搜集。×:必须收集的信息,余为可选收集信息。
- 3、治疗期为PJI治疗手术过程以及术后抗生素使用的过程。×:必须收集的信息,余为可选收集信息。
- 4、随访期V1为手术后抗生素治疗时,若出院后无抗生素治疗计划则在出院时进行V1随访,V2-V6分别定义为抗生素治疗后12周(V2)、24周(V3)、48周(V4)、72周(V5)和96周(V6)。随访方式包括返院复查与远程随访。×:必须收集的信息,余为可选收集信息。
- 5、血常规检查: 白细胞、中性粒细胞计数、血红蛋白、血小板
- 6、炎性指标: 血沉、C 反应蛋白、IL-6(选填)、PCT(选填)、D 二聚体、纤维蛋白原
- 7、血生化检查: ALT、AST、总胆红素、碱性磷酸酶、r-谷氨酰转移酶、总蛋白、白蛋白、尿素 氮、尿酸、肌酐、肌酸激酶、钠、钾、氯、钙、磷、甘油三酯,胆固醇,高密度脂蛋白,低密度 脂蛋白、免疫球蛋白 IgG、血糖。
- 8、 关节液检查: 关节液白细胞计数、中性粒细胞计数及关节液细菌培养

## 附件八:知情同意书

## 临床研究知情同意书

## 尊敬的受试者:

您将被邀请参加一项由福建医科大学附属第一医院张文明主任医师(项目负责人)(电话号码: 13950391800)主持的研究,研究项目名称: 抗生素联合利福平治疗葡萄球菌假体周围感染的疗效与并发症———项多中心、随机对照试验。

您参加本项研究是自愿的,本知情同意书提供给您一些信息以帮助您决定是否参加此项临床研究。本研究已通过福建医科大学附属第一医院伦理委员会审查同意,伦理委员会办公室电话 0591-87981029。如果您同意加入此项研究,请您仔细阅读,如有任何疑问请向负责该项研究的研究者提出。

#### 一、研究目的:

假体周围感染(PJI)是关节置换手术后常见且严重的并发症,给患者带来了巨大的痛苦和治疗挑战。PJI 不仅会延长住院时间,还可能导致手术失败和严重的健康后果。因此,如何有效控制和治疗这种感染成为临床医生关注的重点。在这一过程中,抗生素的使用显得尤为重要,它们是对抗感染的主要武器。

目前,对于 PJI 术后的抗生素治疗方案中是否应添加利福平,以提高感染控制效果,医疗界仍然存在较大分歧。一些研究认为利福平能够增强抗生素的效果,帮助更好地控制感染;而另一些研究则对其具体效果提出质疑,认为需要更多的证据来支持这一做法。由于这些争议,临床实践中对利福平的使用缺乏统一的标准。

为了解决这一问题,我们计划开展一项多中心随机对照临床试验,专门研究联合利福平治疗对 PJI 感染控制的影响。这项研究将汇集多家医院的参与,确保样本的多样性和结果的可靠性。通过严谨的设计和科学的数据分析,我们希望能够明确利福平在 PJI 治疗中的具体作用。

我们的目标是为优化临床抗生素治疗方案提供有力的证据支持,从而帮助医生们在面对 这种复杂感染时做出更好的决策。这不仅有助于改善患者的预后,也为今后的临床治疗提供 了重要的参考依据。

#### 二、研究过程和方法:

如果您同意参与这项研究,我们将为每位受试者分配一个编号,并建立详细的研究档案。本研究将筛选出病原菌为葡萄球菌的 PJI 患者,在经过手术治疗后,静脉使用抗生素治疗 1-2 周后,随机分为利福平联合抗生素治疗组和常规抗生素治疗组,口服抗生素进行为期 3 个月的治疗。在研究期间,患者需要定期复诊,医生将评估感染复发率、炎症指标、假体功能恢复及药物副作用等情况。所有相关数据将被统一记录,并在随访结束后进行分析,以比较两

组在疗效和安全性方面的差异。通过这项研究,我们期望明确利福平联合治疗的效果,从而为 PJI 抗生素治疗方案的优化提供重要依据。

在接受抗生素治疗后的第 1、2、4、6、8、10、12 周,以及 6 个月、9 个月、12 个月、18 个月和 24 个月时,您需要按时回到医院进行复诊,并如实向医生反馈您的病情变化。医生将收集您的病史,并进行常规复查和体检,包括血常规、CRP、ESR、肝肾功能等理化检查。在治疗后的第 24 个月,即出院后 2 年时,研究将结束,您需要再次回到医院进行复诊。医生将询问并记录您的病情变化,并进行体格检查,为您安排必要的血常规、CRP、ESR、肝肾功能等理化检查。

#### 三、研究可能的受益:

参与在本研究您可能不会直接受益,但也有可能因为您的参与,您和社会都会从中获益。 这些潜在的益处包括您的病情可能得到改善,同时本研究可能为 PJI 抗生素治疗方案提供新 的认知,从而帮助类似病情的其他患者。

#### 四、研究风险与不适:

#### 1、服用抗生素所带来的风险:

- 1) 在研究过程中,使用抗生素可能会带来一些副作用。常见的风险包括过敏反应、急性肾功能不全、间质性肾炎等肾功能损害,以及肝功能损害、黄疸、多种血细胞减少、中枢神经系统、消化系统、生殖系统和心血管系统的损害。如果您出现上述任何不良反应,医生将立即停止药物使用,并采取适当的治疗措施,确保您的健康和安全。
- 2) 抗生素可能与其他药物发生相互作用,从而引发副作用。为了您的安全,请在参与本研究前告知医生您正在服用的所有药物,包括处方药、中草药、非处方药、维生素,以及您是否正在接受其他自然疗法或饮用含酒精的饮品等。
  - 3) 耐药菌: 抗生素的使用可能会导致病原微生物产生耐药性, 从而引发耐药菌的出现。。

### 2、可选择的其他诊疗方法:

您有权拒绝参加该研究,或者咨询您的主治医生关于其他常规治疗方法,包括但不限于 喹诺酮类抗生素治疗(例如:环丙沙星、左氧氟沙星、莫西沙星等)。同时,我们也会尽心 为您提供最好的诊疗服务,确保您的健康和安全。

#### 五、隐私问题: (过程中的隐私保护和结果发表的隐私保护)

如果您决定参加本项研究,您参加试验及在试验中的个人资料均属保密。对于您来说, 所有的信息将是保密的。所有的研究成员和研究申办方都被要求对您的身份保密。您的档案 将保存在福建医科大学附属第一医院科研处档案柜中,仅供研究人员查阅。为确保研究按照 规定进行,必要时,政府管理部门或伦理审查委员会的成员按规定可以在研究单位查阅您的 个人资料。该项研究结果发表时,也会对您的身份信息进行保密。

#### 六、费用

如果您选择参与本研究项目,手术期间的诊疗费用以及术后随访的理化检查费用将与您正常接受治疗时产生的费用相同。这些费用是标准医疗过程中的一部分,并不因您参与研究而增加额外费用。在您参与本研究项目的期间,我们将为您提供利福平药物,且不收取任何费用。以下是您的治疗方案详述:

您将被纳入联合抗生素治疗组。在此治疗组中, 您将接受以下药物治疗:

1、常规抗生素治疗,作为基础治疗方案。

2、利福平治疗,作为研究干预措施的一部分,如果您被分配至利福平联合抗生素治疗 组, 您将在常规抗生素治疗基础之上, 额外还需口服利福平, 治疗至满三个月。

利福平的市场单价为 22.93 元人民币, 药品规格为 0.15 克×100 粒。作为本研究的一部 分,您在研究期间使用该药物将不会承担任何费用。

#### 七、补偿

- 1) 研究期间每位患者将给予 1000 元差旅补助费。
- 2) 如果在临床试验中出现不良事件,研究医师将及时采取积极措施进行治疗。

#### 八、自由退出:

作为受试者,您可随时了解与本研究有关的信息资料和研究进展,自愿决定(继续)参 加还是不(继续)参加。参加后,无论是否发生伤害,您可以选择在任何时候通知研究者要 求退出研究,您的数据将不纳入研究结果,您的任何医疗待遇与权益不会因此而受到影响。 在试验过程中,若会对您造成严重的伤害,研究者也将会中止研究的进行。

但在参加研究期间,请您提供有关自身病史和当前身体状况的真实情况;告诉研究医生 自己在本次研究期间所出现的任何不适:不得服用受限制的药物、食物等:告诉研究医生自 己在最近是否曾参与其他研究,或目前正参与其他研究。如果因为您没有遵守研究计划,或 者发生了与研究相关的损伤或者有任何其它原因,研究医师可以终止您继续参与本项研究。

#### 力、联系方式:

如果您有与本研究有关的问题,或您在研究过程中发生了任何不适与损伤,或有关于本 项研究参加者权益方面的问题, 您可以与方心俞医生联系, 电话 18084768503。

#### 十、知情同意签字:

我已经阅读了本知情同意书,并且我的医生 (签字)已经将此次临床试验的目的、内 容、风险和受益情况向我作了详细的解释说明,对我询问的所有问题也给予了解答,我对此 项临床研究已经了解,我自愿参加本项研究。

| 受试者签名: | 研究者签字: |
|--------------------|---------------------|
| 联系手机号: | 联系手机号: |
| 日期: 年月日 | 日期:年月日 |
| (如果受试者不识字时尚需见证人签名, | 如果受试者无行为能力时则需代理人同意) |
| 法定代理人/ 见证人签名: | |
| 与受试者的关系: | |
| 日期: | |

## 附件九:利福平的毒副作用及风险预案

#### 一、 利福平的主要毒副作用

利福平的毒副作用可分为常见和严重两类,在试验中需对副作用进行监测和记录,若

#### 1. 常见副作用(发生率较高,但通常可逆或可管理)

胃肠道反应:恶心、呕吐、食欲不振、腹痛、腹泻。这是**最常见**的不良反应。

体液染色: 汗液、尿液、唾液、泪液等体液呈橘红色。此为正常现象,但需提前告知患者, 避免不必要的恐慌。

肝功能异常:一过性、无症状的肝酶(ALT, AST)轻度升高。

皮肤反应:皮疹、瘙痒。

流感样综合征: 在间歇给药或不规律服药时更常见,表现为发热、寒战、头痛、头晕、骨痛。

#### 2. 严重/罕见副作用(需高度警惕,可能导致停药)

肝毒性:发生情况:可表现为无症状的转氨酶升高,也可进展为肝炎、黄疸,极少数情况下可导致急性肝衰竭。

高危因素: 老年人、原有肝病(如乙肝、丙肝)、酒精滥用、与其他肝毒性药物(如异烟肼) 联用。

血液系统毒性:血小板减少症:可能导致出血倾向。白细胞减少症:增加感染风险。溶血性贫血。

#### 超敏反应:

发生情况:可从轻度皮疹到严重的 Stevens-Johnson 综合征、中毒性表皮坏死松解症等危及生命的反应。

#### 肾毒性:

发生情况:急性间质性肾炎,可导致急性肾损伤。通常与利福平引起的超敏反应有关。 胃肠道严重反应:伪膜性肠炎(由艰难梭菌引起)。

骨骼肌肉系统: 在个别病例中报道有关节痛、肌痛。

#### 3. 特殊的药物相互作用风险(此为利福平最独特的风险之一)

利福平是强效的肝药酶(CYP450系统,特别是CYP3A4)诱导剂,会加速许多药物的代谢,导致其血药浓度下降,药效减弱。这在联合用药时至关重要。

影响本研究核心疗效:需确保联合使用的抗生素(如氟喹诺酮类、夫西地酸等)不与利福平 发生显著的拮抗作用。

#### 影响合并用药:

抗凝药: 华法林效果下降, 增加血栓风险。

心血管药物: 美托洛尔、普萘洛尔、维拉帕米等效果下降。

免疫抑制剂:环孢素、他克莫司血药浓度大幅下降,导致器官移植患者出现排斥反应。

内分泌药物:口服避孕药失效、糖皮质激素、甲状腺激素药效降低。

抗逆转录病毒药:许多HIV药物疗效受影响。

其他: 苯妥英钠、地高辛、茶碱等。

#### 二、 风险预防与应对预案

为确保试验安全,需建立一个贯穿试验始终的、标准化的监测和管理体系,本研究为所有入组的患者购买保险。

#### 预防阶段(试验开始前)

严格的纳入与排除标准。

#### 明确排除:

- 1. 已知对利福平过敏者。
- 2. 活动性、未代偿的肝病患者(如 Child-Pugh B 或 C 级、急性肝炎)、或基线肝功能(ALT/AST) 超过正常值上限(ULN)3倍以上者。
- 3. 严重肾功能不全 (如 eGFR <30 mL/min/1.73m²) 需谨慎。
- 4. 正在使用与利福平有严重相互作用且无法替代或安全调整剂量的药物(见上述药物相互作用列表)。
- 5. 血小板计数、白细胞计数显著低于正常范围者。

全面的基线评估:

- 1. 详细记录患者的既往病史(特别是肝病、酗酒史)。
- 2. 记录所有合并用药,并由研究药师或医生进行药物相互作用筛查。
- 3. 基线检查必须包括:全血细胞计数 (CBC)、肝功能 (ALT, AST, ALP, GGT, 总胆红素)、肾功能 (肌酐, eGFR)、凝血功能 (INR)。

充分的患者知情与教育:

- 1. 签署详细的知情同意书,明确告知利福平的所有常见和严重副作用。
- 2. 特别强调体液变色是正常现象,以及必须规律服药以避免流感样综合征和耐药。
- 3. 教育患者识别严重副作用的迹象(如皮疹、黄疸、异常出血/瘀伤、持续恶心呕吐、深色 尿),并告知出现任何上述症状应立即联系研究人员。

4. 叮嘱患者在看其他疾病或自行购药时,必须告知医生自己正在服用利福平。

#### 监测阶段(试验过程中)

制定标准化的监测时间表(示例):

第1个月:每1-2周复查CBC、肝肾功能。

第2-3个月:每2-4周复查一次。

3个月后:如情况稳定,可延长至每4-8周复查一次。

任何时间点患者报告可疑症状时,立即进行相关检查。

建立严重不良事件(SAE)报告流程:明确各中心的研究者向主要研究者(PI)、伦理委员会和数据安全监察委员会(DSMB)报告 SAE 的时限和路径。

## 应对预案(出现副作用时)

| 副作用类型 | 严重程度 | 处理预案 |
|-------|----------------------|-----------------------|
| | 轻度(无症状,ALT/AST < 3x | 继续用药,加强监测(如1周后复查)。寻找 |
| | ULN) | 其他可能原因(如其他药物、酒精)。 |
| | 中度(ALT/AST 3-5x ULN) | 密切监测,如持续升高或出现症状,考虑暂停 |
| | | 利福平。 |
| 肝毒性 | 重度(ALT/AST >5x ULN, | 立即永久停用利福平。全面评估肝损伤原因, |
| | 或>3x ULN伴黄疸/肝功不 | 给予保肝治疗,直至肝功能恢复。将此事件作 |
| | 全) | 为 SAE 上报。 |
| | 轻度(血小板/白细胞轻度 | 密切监测,每周复查血常规。 |
| | 减少, 无临床症状) | |
| 血液系统毒 | 重度(血小板<50×10°/L, | 立即暂停利福平。评估原因,给予对症支持治 |
| 性 | 或出现出血倾向; 中性粒细 | 疗(如隔离预防感染)。根据恢复情况决定是 |
| | 胞<0.5×10°/L) | 否永久停药。 |
| | 轻度皮疹 | 可考虑使用抗组胺药,并密切观察皮疹变化。 |
| | 严重皮疹(如荨麻疹、水疱、 | 立即永久停用利福平。立即就医,进行紧急处 |
| 超敏反应 | 黏膜受累) 或 SJS/TEN 疑似 | 理。按 SAE 上报。 |
| | | 建议随餐服用(如不影响吸收),或分次服药。 |
| | 轻度恶心/呕吐 | 可使用止吐药。 |
| | | 暂停用药,评估原因(排除伪膜性肠炎),给 |
| 胃肠道反应 | 严重、持续性呕吐/腹泻导 | 予补液支持治疗。待症状缓解后评估是否可重 |
| | 致脱水 | 新尝试给药或永久停药。 |
| | | 首先确认患者是否规律服药。症状严重者需暂 |
| 流感样综合 | 发生 | 停用药,待症状缓解后,可尝试从较小剂量开 |
| 征 | | 始重新给药,并逐步加至全量,或改为每日服 |
| | | 药方案。 |

制定的分级管理策略,所有决定都应由研究者根据患者具体情况做出。

## 关于药物相互作用的预案:

试验前:尽可能调整合并用药,换为不与利福平发生相互作用的药物。

试验中:如需加用新药,必须由研究团队进行相互作用评估,并相应调整剂量(如增加被利福平诱导的药物的剂量),并密切监测其血药浓度(如他克莫司、华法林等)。